CLINICAL TRIAL: NCT06452004
Title: Prevention and Screening Intervention Project - Towards Elimination of Cervical Cancer: Validation of Artificial Intelligence as Decision Support System in VIA
Brief Title: Validation of Artificial Intelligence as Decision Support System in VIA (PRESCRIP-TEC)
Acronym: AI-DSS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Uganda Cancer Institute (Other); Female Cancer Foundation (Unknown); International Centre for Diarrhoeal Disease Research, Bangladesh (Other); Manipal Academy for Higher Education (Unknown); Friendship Bangladesh (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2022300195
Record Dates: First submitted 2023-10-26; First posted 2024-06-11 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2024-06

CONDITIONS: HPV Infection; Cervix Cancer; Cervical Dysplasia
Keywords: Visual Inspection cervix; Artificial Intelligence; Screening Cervical Cancer; decision support system
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms; Uterine Cervical Dysplasia

STUDY DESIGN:
Intervention Model Description: In Uganda, India and Bangladesh eligible women in geographic areas are invited to perform self-test for hrHPV. hrHPV-positive women are invited for further examination of the cervix using VIA. In all VIAs pictures are taken with the device and the AI decision support system is activated. Health workers will give an independent VIA assessment before the AI assessment can be accessed. An expert panel gives an independent assessment without knowing the health worker or AI assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- AI-DSS validation Bangladesh (Experimental): Women in selected intervention area in Bangladesh, who tested hrHPV-positive eligible for VIA, are included. VIA is performed. During VIA the health worker performs an assessment. With the device a picture and taken and AI-DSS generates and assessment as well. The pictures are also assessed by an expert panel.
  Interventions: Diagnostic Test: Validation of AI-DSS in Bangladesh
- AI-DSS validation Uganda (Experimental): Women in selected intervention area in Uganda, who tested hrHPV-positive eligible for VIA, are included. VIA is performed. During VIA the health worker performs an assessment. With the device a picture and taken and AI-DSS generates and assessment as well. The pictures are also assessed by an expert panel.
  Interventions: Diagnostic Test: Validation of AI-DSS in Uganda
- AI-DSS validation India (Experimental): Women in selected intervention area in India, who tested hrHPV-positive eligible for VIA, are included. VIA is performed. During VIA the health worker performs an assessment. With the device a picture and taken and AI-DSS generates and assessment as well. The pictures are also assessed by an expert panel.
  Interventions: Diagnostic Test: Validation of AI-DSS in India

INTERVENTIONS:
Diagnostic Test: Validation of AI-DSS in Bangladesh — VIA procedure, taking pre-colouring and post-colouring pictures. First VIA assessment by health worker, followed by AI-DSS assessment. Independent panel of gynaecologists also assessed pictures. The panel assessment serves as reference value to calculate accuracy, sensitivity and specificity of health worker and AI-DSS.
  Arms: AI-DSS validation Bangladesh
Diagnostic Test: Validation of AI-DSS in Uganda — VIA procedure, taking pre-colouring and post-colouring pictures. First VIA assessment by health worker, followed by AI-DSS assessment. Independent panel of gynaecologists also assessed pictures. The panel assessment serves as reference value to calculate accuracy, sensitivity and specificity of health worker and AI-DSS.
  Arms: AI-DSS validation Uganda
Diagnostic Test: Validation of AI-DSS in India — VIA procedure, taking pre-colouring and post-colouring pictures. First VIA assessment by health worker, followed by AI-DSS assessment. Independent panel of gynaecologists also assessed pictures. The panel assessment serves as reference value to calculate accuracy, sensitivity and specificity of health worker and AI-DSS.
  Arms: AI-DSS validation India

SUMMARY:
The research project is a component of another research project that applies the protocol of the World Health Organization for screening of cervical cancer, with testing of high-risk Human Papilloma Virus (hrHPV) as first screening. In the screen, triage and treat approach women who tested positive for hrHPV are undergoing Visual Inspection of the cervix with Acetic Acid (VIA). This procedure is applied in Uganda, India and Bangladesh. However the quality of VIA by lower-trained staff is variable because Low and Middle Income Countries face limited numbers of qualified health care professionals. Artificial intelligence (AI) might be a solution to improve consistency of VIA assessment. This research validates an AI decision support system (AI-DSS) under field conditions.

DETAILED DESCRIPTION:
This research project aims to validate an image processing algorithm in order to study if the AI can function as decision support system (DSS) for healthcare workers, who perform VIA. The AI-DSS has been designed by the Manipal Academy of Higher Education in India and has shown a sensitivity of 99.05% and specificity of 97.16% for detection of aceto-white lesions.

The first step of the validation process is a dry run using a database of VIA pictures with pathology confirmation. The accuracy, sensitivity and specificity of healthcare workers, an expert team and the AI will be analysed, based on the ground truth of database pictures.

Thereafter, the AI-DSS will be validated under field conditions. Women who are hrHPV-positive in Uganda, India and Bangladesh will undergo a VIA. The AI is incorporated in a device, that can take pictures of the cervix and provide and instant report (positive = needs further investigation or negative = no lesions found). The user experience of the device will be evaluated.

The AI-DSS will be validated by comparing the VIA assessment by health workers, the AI with assessment by the expert panel. Accuracy, sensitivity and specificity of the AI algorithm will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Female in eligible age group
* Women who tested HPV positive and are eligible for VIA
* Ability to give informed consent and participate in study

Exclusion Criteria:

* Clinical signs of cervical carcinoma
* Menstruation or other vaginal blood loss
* HPV negative women

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 600 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy, sensitivity, specificity of AI-DSS | through study completion, estimated 2 years
  Measurement of true and false positive and true and false negative results of the AI DSS in relation to assessment by expert panel

SECONDARY OUTCOMES:
Percentage of quality pictures | through study completion, estimated 2 years
  Percentage of pictures taken during the VIA procedures, which meet according to the expert panel the quality standards suitable for AI-DSS assessment, based on visibility of cervix and Squamo-Columnar Junction (SCJ), light, reflection of speculum, mucus-free surface

OTHER OUTCOMES:
User-friendliness of AI-DSS device among healthcare providers | through study completion, estimated 2 years
  Scoring on Likert scale by healthcare providers using AI-DSS device based on their assessment of device software human machine interface, weight, size, flashlight,

CONTACTS AND LOCATIONS:
Overall Officials: Jelle Stekelenburg, MD, PhD, Principal Investigator — University Medical Center Groningen; Janine de Zeeuw, PhD, Principal Investigator — University Medical Center Groningen; Jogchum Beltman, MD, PhD, Principal Investigator — Female Cancer Foundation; Keerthana Prasad, PhD, Principal Investigator — Manipal Academy for Higher Education; Carol Nakisige, MD, Principal Investigator — Uganda Cancer Institute; Aminur Rahman Shaheen, PhD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- Mpasana, Kakumiro, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Sharing according to the European Union Open Research guidelines
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After 1 January 2024
Access Criteria: As per Open Research Protocol, on request to Principal Investigator UMCG
URL: http://www.prescriptec.org

REFERENCES:
- [Background] Sultanov M, Zeeuw J, Koot J, der Schans JV, Beltman JJ, Fouw M, Majdan M, Rusnak M, Nazrul N, Rahman A, Nakisige C, Rao AP, Prasad K, Guruvare S, Biesma R, Versluis M, de Bock GH, Stekelenburg J. Investigating feasibility of 2021 WHO protocol for cervical cancer screening in underscreened populations: PREvention and SCReening Innovation Project Toward Elimination of Cervical Cancer (PRESCRIP-TEC). BMC Public Health. 2022 Jul 15;22(1):1356. doi: 10.1186/s12889-022-13488-z. PMID 35840949
- [Background] Nakisige C, de Fouw M, Kabukye J, Sultanov M, Nazrui N, Rahman A, de Zeeuw J, Koot J, Rao AP, Prasad K, Shyamala G, Siddharta P, Stekelenburg J, Beltman JJ. Artificial intelligence and visual inspection in cervical cancer screening. Int J Gynecol Cancer. 2023 Oct 2;33(10):1515-1521. doi: 10.1136/ijgc-2023-004397. PMID 37666527